CLINICAL TRIAL: NCT04022382
Title: A Single-Arm, Single-Center, Randomized, Single-Masked Study to Evaluate Restylane-Defyne for Punctal Occlusion in Participants With Mild to Moderate Dry Eye Disease
Brief Title: A Study to Evaluate the Safety and Effectiveness Assessments of Restylane-Defyne for Punctual Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John C Meyer, MD (Other)
Responsible Party: Sponsor-Investigator, John C Meyer, MD, Ophthalmologist, The Eye Care Institute
Organization: The Eye Care Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0619
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Dry Eye
Keywords: Dry Eye Disease; Restylane-Defyne
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Restylane Defyne recipient (Experimental)
  Interventions: Device: Restylane Defyne

INTERVENTIONS:
Device: Restylane Defyne — Restylane is a gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL.

SUMMARY:
A study which participants with mild to moderate dry eye disease will have a punctum of one eye injected with 0.1ml Restylane Defyne and the other eye injected with 0.2ml Restylane Defyne. Participants will be evaluated over four visits.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 80 years of age
* Baseline OSDI score of at least 13 with no more than 3 responses of "not applicable"
* In both eyes, a baseline Schirmer test with anesthetic of ≤ 10mm/5 minutes
* Literate, able to speak English and able to complete the questionnaire independently
* Willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol.

Exclusion Criteria:

* Use of ophthalmic cyclosporine or lifitegrast within 30 days prior to Day 0
* History of surgical punctal occlusion (e.g., cautery), canalicular infection or canalicular surgery
* Corneal transplant in either eye
* Ocular surgery (such as cataract surgery or LASIK) in either eye within six months of the Baseline Visit
* A systemic condition or disease not stabilized or judged by the investigator to be incompatible with participation in the study (e.g. current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease)
* The history or presence of any ocular disorder or condition in either eye that, in the opinion of the investigator, would interfere with the interpretation of the study results (e.g., significant corneal or conjunctival scarring, pterygium or nodular pinguecula; current ocular infection (except mild blepharitis), conjunctivitis or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; history of ocular herpetic infection; evidence of keratoconus; lid or lacrimal cancer.
* Active severe systemic allergy, seasonal allergies, rhinitis or sinusitis requiring changes in treatment within 30 days prior to the study or likely to require changes in treatment during the course of the study (i.e. antihistamines, decongestants, oral, topical or aerosol steroids)
* Participation in a clinical trial during the past 30 days
* Women who are pregnant, planning a pregnancy, or nursing at study entry.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Evaluating change in Schirmer score from baseline. | 30 days
  Maximum length of tears absorbed on test strips recorded.

SECONDARY OUTCOMES:
Evaluating change in OSDI score. | 30 Days
  Participants answer 12 question questionnaire. Scores from section I,II, and III.
Evaluating change in corneal staining score. | 30 Days
  1.0mg sodium fluorescein strips on lower eye lids for one minute. 5 corneal regions graded using cobalt filter to maximized view of fluorescence.
Evaluating change in dye disappearance test. | 30 days
Evaluating change in tear break-up time. | 30 days
  Performed by Keratograph 5M per manufacturer's directions.
Evaluating change in tear meniscus height. | 30 days
  Performed by Keratograph 5M per manufacturer's directions.

CONTACTS AND LOCATIONS:
Overall Officials: John C Meyer, MD, Principal Investigator — The Eye Care Institute
Locations (1):
- The Eye Care Institute, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No